CLINICAL TRIAL: NCT04447196
Title: Prevalence of Rest Dyspnea and Impact of Non Invasive Ventilation on Breathing Sensations in Patients With Congenital Central Hypoventilation Syndrome
Brief Title: Prevalence of Rest Dyspnea and Impact of Non Invasive Ventilation on Breathing Sensations in CCHS Patients
Acronym: DyspnOndine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00215-34
Record Dates: First submitted 2020-05-30; First posted 2020-06-25 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: CCHS; Congenital Central Hypoventilation Syndrome; Dyspnea
MeSH Terms: conditions — Congenital central hypoventilation syndrome; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCHS: 20 patients presenting with central hypoventilation syndrome during spontaneous breathing and with Non Invasive Ventilation
  Interventions: Other: MDP

INTERVENTIONS:
Other: MDP — Multi dimensional dyspnea profile scores at rest and during non invasive ventilation

SUMMARY:
Congenital central hypoventilation syndrome (CCHS) is a neuro-respiratory disease characterized by lifethreatening sleep-related hypoventilation involving an alteration of CO2/H+ chemosensitivity. This suggests cortical activity during awakening to maintain breathing. Cortical activity to keep breathing is usually associated with breathing discomfort ; this is the case in healthy subjects under non invasive ventilation (NIV) or with expiratory charge as well as in patients with amyotrophic lateral sclerosis. This can suggest that CCHS may be breathless at rest and this discomfort could be reduced by NIV.

The objective is to evaluate dyspnea with a multi dimensional score, MDP, in CCHS patient at rest in every day life and during 1H session of NIV.

The investigators will perform a prospective, including 20 CCHS patients. MDP scores will be measure before and after 1H-non invasive ventilation as well as a visual scale of 100mm in order to evaluate variation of breathing discomfort before/after NIV.

The investigators expect that CCHS patients don't have rest dyspnea but NIV would improve breathing discomfort that would mean they have latent rest dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* patients with CCHS confirmed by genetic test
* patients with long term non invasive ventilation
* no recent condition that could impact breathing sensations such as infection, pulmonary embolism, heart failure

Exclusion Criteria:

* pregnancy
* phrenic nerve stimulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with CCHS who already require long terme NIV but not phrenic nerve stimulation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
"Immediate unpleasantness" corresponding to A.1 item of the multidimensional dyspnea profile | Change in MDP score between baseline and after 1 hour of NIV
  Measure MDP scores before and after NIV

CONTACTS AND LOCATIONS:
Locations (1):
- INSERM-UPC UMR_S 1158, Service de Pneumologie et Réanimation, GH Pitié-Salpêtrière, Paris, France